CLINICAL TRIAL: NCT00418704
Title: A Multicenter Randomized Phase II Trial in NSCLC Stage IV and IIIB (T4 With Pleural Effusion) in Elderly Independent Patients the Schedule Docetaxel / Gemcitabine First Line Following by Erlotinib When Progression Versus Erlotinib First Line Following by/ Gemcitabine When Progression.
Brief Title: Elderly Independent Patients With Non Small Cell Lung Cancer (NSCLC)
Status: Completed | Type: Observational
Sponsor: Groupe Francais De Pneumo-Cancerologie (Other)
Collaborators: Sanofi (Industry); Chugai Pharma USA (Industry)
Responsible Party: Sponsor
Other Study IDs: GFPC 05-04
Record Dates: First submitted 2007-01-04; First posted 2007-01-05 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: cancer; Lung cancer; None small-cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Lung Neoplasms | interventions — Erlotinib Hydrochloride; Docetaxel

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Erlotinib — Tarceva (150 mg) is a pill you take once a day -- every day
Drug: taxotere — Taxotere® (docetaxel) is given intravenously (I.V.) into the vein. Taxotere® chemotherapy treatment takes about one hour, and usually people receive treatments every three weeks.
  Other Names: Docetaxel

SUMMARY:
The purpose of this study is to determine duration before progression of first-line treatment chemotherapy following erlotinib in second-line comparing erlotinib in first-line following chemotherapy in second-line in old patients with none small cell lung cancer.

DETAILED DESCRIPTION:
A multicenter phase II trial , prospective, randomized, open, non comparative

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 years
* Comorbidities score,
* PS frailty score**.according to(TABLE N°1)
* No dementia, repeated falls, faecal or urinary incontinence, ADL=0, IADL=0
* Life expectancy at least 12 weeks
* Créatinine clearance de la créatinine > or =30cc/mn according to Cockrofts
* Gault formula
* Competency to give written informed consent
* Haematological function as follows: absolute neutrophil count > 1.5 x 109/l and/or platelet> 100 x 109/l, hémoglobine > or = 9,5 g/dl
* Hepatic function as followed :bilirubin <1,25 LNS SGOT/SGPT <5 x N,PAL <5N
* PS < 3
* No symptomatic cerebral metastasis
* Histologically or cytologically confirmed NSCLC
* Stage IV/IIIB4 (T4with pleural effusion)
* No prior chemotherapy for NSCLC
* Relapses of previous NSCLC treated by surgery or radiotherapy are eligible if the target is measurable out of initial radiotherapy field and if histological or cytological proof
* At least one measurable target lesion by RECIST guidelines.

Exclusion Criteria:

* Symptomatic cerebral metastasis
* Any severe co-morbidity calculated by Charlson score (according to table 1), any kind of disorder that compromises the ability of the subject to give written informed and/or comply with the study procedure ADL > or = 1 et IADL > or =1 Dementia, repeated falls, faecal or urinary incontinence- Peripheral neuropathy grade 2 or more
* Performance Status > 2 ( ECOG)- Contraindication to corticosteroids
* Unwilling or unable to comply with study requirements for personal , family, sociologic, geographic or any reasons
* Lack of liberty following administrative or judicial decision
* Hypersensitivity to polysorbate
* Hypersensitivity to erlotinib or any excipients of this product
* Unusual hereditary disorders as galactosemia, deficit in lactase and malabsorption in glucose or galactose
* Participation in concomitant clinical trial
* Contraindication to a product of this study disease
* Bronchioloalvéolar or neuroendocrine or composite carcinoma
* Superior vena cava syndrome

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with non small-cell lung cancer stage IV and IIIB (T4 with pleural effusion) in elderly independent patients évaluant
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2006-05; Primary Completion 2006-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hervé LECAER, Doctor, Principal Investigator — Groupe Francais De Pneumo-Cancerologie
Locations (22):
- France (22):
  - Site 12, Aix-en-Provence
  - Site 22, Beauvais
  - Site 30, Charleville-Mézières
  - Site 48, Clermont-Ferrand
  - Site 33, Créteil
  - Site 07, Draguignan
  - Site 32, Elbeuf
  - Site 04, Gap
  - Site 41, Le Chesnay
  - Site 00, Limoges
  - Site 25, Mantes-la-Jolie
  - Site 06, Marseille
  - Site 27, Martigues
  - Site 01, Meaux
  - Site 26, Paris
  - Site 19, Périgueux
  - Site 02, Reims
  - Site 20, Rennes
  - Site 18, Rouen
  - Site 17, Rouen
  - Site 14, Toulon
  - Site 11, Villefranche-sur-Saône

REFERENCES:
- See also: Groupement Francais de Pneumo-cancérologie — http://www.g-f-p-c.org